CLINICAL TRIAL: NCT07386652
Title: Randomised Controlled Trial of an Intensive Comprehensive Aphasia Programme for People With Post-Stroke Aphasia
Acronym: RCT of an ICAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 177373
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Aphasia Following Cerebral Infarction
Keywords: Intensive Comprehensive Aphasia Programme; ICAP; People With Aphasia; PWA
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Comprehensive Aphasia Programme (Experimental): As defined by the new framework commissioned by the NIHR and the MRC [44], ICAPs are complex interventions with multiple interacting components. We have published our ICAP operating manual using the TIDieR format (Template for Intervention Description and Replication) to ensure it complies with intentionally accepted requirements (see uploads) [45, 46] Accordingly, no individual PWA or their carer will receive all possible therapeutic components; instead, the therapists will personalise content according to individual needs to help them achieve their goals. A further key feature of the ICAP is that the treating therapists (4 Speech and Language Therapists and one Clinical Psychologist) work as a team, meaning all of them will work with each PWA over the 4-week ICAP.
  Interventions: Behavioral: ICAP
- Control (standard care) (Active Comparator): Although the amount of therapy received by PWA in the community varies, the most in-depth study of this variation across 21 UK-based SLT departments concludes as follows: "Where resources are in short supply, therapists have the difficult ethical decision of providing therapeutic levels of intervention to some patients, or providing sub therapeutic levels to all. Currently it looks as if the latter is most common in practice."[48] This study found the majority of PWA over a year post-stroke were not receiving any therapy, while a minority were receiving ~6.3 hours, ranging widely from 0.5-41.5 hours. To capture the quantity and quality of the therapy received by PWA in this arm (and the ICAP group once they complete the ICAP) we will ensure the research team complete the relevant sections of the Client Service Receipt Inventory at each time point
  Interventions: Behavioral: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: ICAP — As defined by the new framework commissioned by the NIHR and the MRC [44], ICAPs are complex interventions with multiple interacting components. We have published our ICAP operating manual using the TIDieR format (Template for Intervention Description and Replication) to ensure it complies with intentionally accepted requirements (see uploads) [45, 46] Accordingly, no individual PWA or their carer will receive all possible therapeutic components; instead the therapists will personalise content according to individual needs to help them achieve their goals. A further key feature of the ICAP is that the treating therapists (4 Speech and Language Therapists and one Clinical Psychologist) work as a team, meaning all of them will work with each PWA over the 4-week ICAP.
  Arms: Intensive Comprehensive Aphasia Programme
Behavioral: Standard Care (in control arm) — Although the amount of therapy received by PWA in the community varies, the most in-depth study of this variation across 21 UK-based SLT departments concludes as follows: "Where resources are in short supply, therapists have the difficult ethical decision of providing therapeutic levels of intervention to some patients, or providing sub therapeutic levels to all. Currently it looks as if the latter is most common in practice."[48] This study found the majority of PWA over a year post-stroke were not receiving any therapy, while a minority were receiving ~6.3 hours, ranging widely from 0.5-41.5 hours. To capture the quantity and quality of the therapy received by PWA in this arm (and the ICAP group once they complete the ICAP) we will ensure the research team complete the relevant sections of the Client Service Receipt Inventory at each time point.
  Arms: Control (standard care)

SUMMARY:
Research question Does participation in an Intensive Comprehensive Aphasia Programme produce a meaningful change in the communication of people with aphasia, their quality of life and that of their carers?

Background Aphasia is a persistent language disorder that severely impairs communicative abilities. Most commonly induced by a stroke, aphasia reduces quality of life more than any other condition. People with aphasia (PWA) and their carers feel abandoned by the NHS due to the limited treatment options available. Meanwhile, neuroscientific evidence suggests that PWA can make meaningful gains in communicative ability, mood, and quality of life if therapists are given enough time to work with them. Although studies indicate Intensive Comprehensive Aphasia Programmes (ICAPs) are effective ways to deliver such therapy, no randomised controlled trial (RCT) of an ICAP has yet been conducted. We propose conducting the first ever ICAP RCT.

Aims and objectives Clinical: i) To test the efficacy of an ICAP in improving PWAs' language impairment, communicative ability, mood, and quality of life; ii) to measure the quantity and quality of therapy received in the community by the standard care group; iii) to assess the significance of age and time-since-stroke in PWA's responses to ICAP intervention.

Mechanistic: To test whether combining baseline behaviour and MRI brain scans can usefully predict individual patients' responses to the ICAP treatment.

Methods Our RCT will test the effect of an ICAP intervention by randomly assigning PWA and their carers to one of two groups receiving either ICAP or standard care at two participating sites. We aim to deliver 100 hours of ICAP therapy over a 4-week schedule to adult PWA who are more than 3 months post-stroke. We will compare the effects of the ICAP, comprising complex interventions with multiple interacting therapeutic components, with standard care, the quantity and quality of which will be recorded by research assistants. The primary outcome measure is a standardized scale for measuring quality of life for PWA (SAQOL-39g). The primary endpoint is 4 months post-randomisation. We will also test for effects at 9 months.

Anticipated impacts Our trial could provide the evidence needed to transform how the NHS treats PWA and their carers. If we demonstrate that participating in an ICAP leads to clinically meaningful and sustained improvements, the next stage in achieving wider NHS roll-out will be a multi-centre trial to investigate the cost- and clinical effectiveness of ICAPs across the UK.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Why is this research needed now? Aphasia is a distressing and increasingly prevalent condition Aphasia is an acquired disorder of language that often persists as a lifelong condition following a brain injury. A stroke is by far the commonest cause, with aphasia experienced by a third of stroke survivors.

In a study of over 66,000 people dependent on others for care, aphasia was rated worse than 75 conditions associated with poor quality of life, including cancer, dementia, quadriplegia, and motor-neurone-disease [1].

The Stroke Association estimates 350,000 people have post-stroke aphasia in the UK, and this number is set to increase significantly. Although new cases of stroke in high-income countries are decreasing by around 1% per year across all age bands [2], the aging populations of these countries mean the number of people living with stroke will double by 2035. The prevalence of PWA will thus rise despite the lower incidence of strokes.

While acute stroke services have been transformed by the use of thrombolysis and thrombectomy to reduce disability, only 10% of people are currently able to receive thrombolysis and 2% are able to receive thrombectomy in the UK [3]. Meanwhile, the number of people surviving strokes with life-changing language impairments is set to increase for at least the next 30 years [4].

Effective speech and language rehabilitation has an increasingly important role to play at a time when the numbers of PWA are rising and receiving ever-fewer resources.

Aphasia not only adversely affects PWA but all those in their social circle, primarily because it reduces a person's ability to connect with others. Aphasia has especially negative impacts on family members and loved ones, who often become the de facto carers of PWA [5]. Yet carers get even less support in dealing with these impacts than PWA, leaving them feeling emotionally distressed, trapped, burdened, unable to work, and 'burned out' [6].

Current speech and language therapy approaches are effective but PWA remain massively under-dosed The good news is PWA can make significant gains in their communicative abilities even years after a stroke. Crucially, however, such gains require many hours of guided practice. Unfortunately, PWA continue to get only 4 hours of speech and language therapy (SLT) as in-patients (3) and 8 SLT sessions in the community [7], amounting to roughly 10% of the dose needed to make meaningful improvements in their communicative abilities [8, 9].

This critical under-dosage persists despite NICE having recently changed its guidelines to call for an increase in the hours and intensity of speech therapy for PWA [10] and despite the National Clinical Guidelines for Stroke now recommending speech therapy be offered for as long as PWA continue to benefit [11].

Evidence from meta-analyses of interventional studies on PWA confirms the importance of sufficient therapy dose for achieving clinically meaningful change: Bhogal's seminal meta-analysis suggested 100 hours [8]; the latest Cochrane review suggests 60-208 hours [12]; and the most recent evidence from the RELEASE project indicates that 3-5 days of therapy per week leads to the greatest gains in overall language and functional communication [9].

Given this evidence, the challenge is how to deliver sufficiently high doses of contact with expert coaches (therapists) to make a difference to PWA. Although evidence from some aphasia studies supports theoretical claims that spacing out therapy may be beneficial [13], economic factors have driven a rise in intensive programmes (ICAPs) as a way of providing large doses over short time scales. This is essentially because therapy teams working at single sites are more efficient than peripatetic solo therapists.

The aim of ICAPs is to produce a step-change in language function sufficient to enable PWA to engage more effectively with others and to continue to maintain and even boost any ICAP-related gains in communication.

The minimum number of contact hours for a service to be considered an ICAP is 3 hours a day for two weeks [14], i.e. >30 hours in total, which is far more than most community-based PWA ever receive [15]. To date, 9 ICAPs that have treated 10 or more PWA have published their findings, with each employing a pre-post analysis using a variety of standardised outcome measures. Table 1 (below) summarises the key attributes of these ICAPs, including effect sizes on impairment and function-based outcome measures. In sum, most have demonstrated medium to large effects on key language impairment and functional outcome measures [16, 17].

Aphasic strokes affect many aspects of people's lives; this ICAP will target the 4 key ones Post-stroke aphasia has multiple adverse effects. Compared with age-matched controls and people with left-hemisphere strokes but no aphasia, people with persistent aphasia caused by a stroke have a higher incidence of associated non-language cognitive impairments [18]. These primary impairments (shaded blue in Figure 1) have secondary effects (shaded orange), including social isolation [19] and low mood, with depression affecting 43-70% of PWA [20]. Indeed, PWA are 7 times more likely to suffer from depression than people who have had a stroke but no aphasia [21]. Together these primary and secondary effects have knock-on negative impacts on PWA's quality of life [22]. Our ICAP model will target all 4 effects through specific interventions delivered by trained therapists (depicted in Fig 1 by green people icons). The ultimate aim of these interventions is to make meaningful improvements in the quality of life of PWA and their carers. This goal reflects the declared priorities of PWA and their family members [23].

Carers count too! The ICAP will specifically target carers of PWA Over half of all PWA depend on support from carers for everyday activities and emotional health. Most carers are spouses, family members, or other close contacts of PWA. Caring for PWA is strongly associated with emotional distress and feeling overburdened.

Carers have little time to adjust to their loved ones losing their pre-stroke identity and the changes in roles arising from dependency. Negative outcomes are common among caregivers in the first months after stroke onset and tend to persist for months and even years. Rates of depression of 11- 42% have been reported among carers [24]. Depression, stress, poor family functioning and other caregiver-related factors also correlate with negative outcomes for stroke survivors, including their rates of functional recovery and stress [25].

"It feels as though the majority of responsibility for recovery falls on me." (Parent of Year 2 Queen Square ICAP participant)

What are ICAPs and why might they be effective? ICAPs offer high-dose and high-intensity face-to-face therapy to PWA and their carers. Internationally accepted guidelines define the minimum measures constituting adequate ICAP services, including the minimum dose (30 hrs) and intensity (3 hrs per day) of aphasia treatment. This therapy should be delivered in group contexts so PWA can learn from each other [26]. Since ICAPs are complex interventions that target the main 3 areas of the WHO International Classification of Functioning, Disability and Health (ICF), they are necessarily holistic. And since they involve carers, they are also systemic. Despite such complexity, ICAPs can be understood simply as providing therapists the time and space needed to deliver effective doses of interventions they are already trained to perform.

OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS Aims

We will address 3 key gaps in the current evidence base that need resolving before wider implementation of ICAPs can proceed:

1. We will conduct the first ever RCT of an ICAP to test if the clinical effect sizes are as large as observational studies have reported. If ICAPs are to be rolled-out in the NHS, we need to demonstrate what the true effect sizes are by comparing the ICAP with a matched sample of PWA undergoing standard care (reflecting current practices).
2. We will carry out secondary analyses to see if two key PWA variables significantly affect the main result: 1) the age of PWA and 2) time-since-stroke. This will help personalise ICAP provision if either or both variables prove important modulators of therapy effects.
3. By using a high-resolution MRI brain scan prior to therapy, we will provide a mechanistic account of the effects of the ICAP on PWA's speech production and speech comprehension gains. This will enable future stratification of PWAs based on brain imaging.

Clinical Objectives

1. To test whether an ICAP produces a clinically meaningful improvement in PWA's language impairment, communicative ability, mood and quality of life compared with standard care.
2. To measure the quantity and types of intervention that PWA receive in the community (both groups).
3. To investigate whether age and time-since-stroke are significant factors in determining PWAs' response to an ICAP.

Mechanistic Objectives

1. To test whether individual responses to ICAP treatment are predictable, i.e. whether we can best predict individual outcomes based on a person's baseline behaviour and MRI brain scan.
2. To test whether ICAP-driven improvements in language production and comprehension among individual PWA depend on the intactness of different brain regions.

3.1 Primary Objectives

Clinical (key quantitative hypotheses tested using between-group comparisons):

Compared with standard care, does an ICAP intervention result in statistically significant and clinically meaningful improvements for PWA at 4 months in the following key domain?

a. Quality of life, as measured by the Stroke and Aphasia Quality of Life Scale-39 [27]

Mechanistic (to be achieved by combining brain imaging data and behavioural data from PWA randomised to the ICAP):

Can we predict individual responses of PWA to ICAP therapy based on their baseline behaviour and structural MRI brain scan?

Secondary Objectives Clinical

1. Compared with standard care, does an ICAP intervention result in statistically significant and clinically meaningful improvements for PWA at 4 months in the following key domains?

   1. Language impairment, as measured by the Comprehensive Aphasia Test [28]
   2. Communication, as measured by the carer-rated Communicative Effectiveness Index [29]
   3. Confidence, as measured by the Communication Confidence Rating Scale for Aphasia [30]
   4. Mood, as measured by the Stroke Aphasic Depression Questionnaire [31]
   5. Carer burden, as measured by the Adult Carers Quality Of Life Questionnaire [32]
2. Does time-since-stroke or age significantly affect ICAP-induced effects on any of the outcome measures mentioned above?

   Mechanistic
3. Are ICAP-driven improvements in language production and comprehension dependent on damage to/intactness of different brain regions? We will test whether:

   1. Improvements in comprehension skills are significantly greater when the cerebellum, supramarginal gyrus and superior temporal cortex are preserved. All 3 regions are known to play a role in receptive language [33, 34], and damage in these areas was also strongly correlated with the gains patients made in their receptive language skills during the Queen Square ICAP (Fig 5).
   2. Improvements in speech production are significantly greater when the Rolandic operculum, the middle frontal gyrus and the cingulum are spared. The Rolandic operculum is well known to play a role in normal speech production [35]. Although the middle frontal gyrus and cingulum are less obviously prominent in speech [36], their destruction might interfere with broader sensory-motor integration functions, which in turn hamper patients' ability to respond to ICAP treatments.
   3. Notably, the regions for predicting improvement in language comprehension are all involved in the same function in the premorbid brain. However, the regions predicting improvement in language production also include those involved in more general cognitive domains (Fig 5). This suggests that different mechanisms of recovery are at play for two of the key language domains. We will test if this pattern is consistent in the larger sample.

TRIAL DESIGN The ICAP will be evaluated as a 2-arm group RCT across two sites: North London (Queen Square) and South London (St. George's). The comparator will be 'standard care', the quantity and quality of which will be recorded using the Client Service Receipt Inventory [37].

Allocation to these groups will be on a 1:1 ratio. To ensure the groups do not become unbalanced we will use stratified randomisation based on two factors: aphasia severity and time-since-stroke. The allocation will be balanced at each site and will be carried out by the Bangor Clinical Trials Unit.

SAMPLING METHODS Study population We want to ensure that our sample population (i.e. the PWA who enter the trial) is as representative as possible of our study population, which is all PWA with access to the NHS. Although we only have two sites (as this is an efficacy study), by basing them in London we hope to include PWA from diverse ethnicities, particularly at the St George's site. Since the Queen Square site is a national referral centre, we will also capture regional diversity (see the map and recruitment section below for more details). For the previous Queen Square ICAP, 50% of those assessed in a general aphasia assessment clinic were deemed eligible.

Withdrawal criteria: those PWA unable to tolerate the ICAP dose/intensity (defined as completing less than 50% of the planned sessions across the 4 weeks). In the two years of the Queen Square ICAP, only one of the 90 participants dropped out.

Inclusion criteria

1. Adult (>18 years old) PWA caused by stroke
2. More than 3 months post-stroke
3. Can use English to communicate (even if not as their first language)
4. Carers will be nominated (if available) by individual PWA

Exclusion criteria

1. Severe speech apraxia (no meaningful spoken word output)
2. Severe fatigue or other reasons they cannot commit to the timing and duration of the ICAP
3. Ongoing debilitating psychiatric disorders (e.g. psychosis, but not low mood)
4. Co-existing neurological disorders affecting engagement (e.g. dementia).

Recruitment Recruitment method and consent process Consistent with our multifaceted recruitment approach to promote ethnic, linguistic, and social diversity in our trial, we will recruit participants through two diverse NHS sites and voluntary sector and community groups more broadly. Our study processes are designed to address logistical barriers, including transport costs associated with trial participation.

Having previously published studies that successfully recruited from areas with high socio-economic deprivation, we appreciate some communities are more hesitant to take part in research. Accordingly, we will use evidence-based approaches such as staff cultural competence training, recruitment videos in Languages Other Than English (LOTE) and leverage community partnerships to build rapport and apply a personalised approach [38]. We will work closely with our advisory groups and local clinicians on how best to widen access, e.g. by involving Community Support workers and other trusted members of local communities.

Overview of research methods to capture data from participants and their frequency Participants will complete questionnaires and tests to capture demographic, case history and outcome measures at baseline, 1 month (post-intervention), 4 months, and 9 month (follow-up). The study researchers collecting data will be speech and language therapists experienced in working with PWA.

Informed Consent Type and content of participant information materials Participant information sheets (PIS) and consent forms will be developed applying aphasia-accessible principles (e.g. using short simple sentences, presenting key ideas with suitable pictorial images, emboldening key words) [42]. The PIS will also be developed as a video for those who find it difficult accessing written information [39]. To facilitate inclusion of those who speak English as an additional language, the information videos, PIS and consent forms will be translated in the 3 most common LOTE identified through our sites and PPI. We will take advice from sites and advisory groups on making patient-facing documents and videos sensitive to different cultures, backgrounds, and identities.

INTERVENTIONS Experimental intervention (ICAP) As defined by the new framework commissioned by the NIHR and the MRC [44], ICAPs are complex interventions with multiple interacting components. We have published our ICAP operating manual using the TIDieR format (Template for Intervention Description and Replication) to ensure it complies with intentionally accepted requirements (see uploads) [45, 46] Accordingly, no individual PWA or their carer will receive all possible therapeutic components; instead the therapists will personalise content according to individual needs to help them achieve their goals. A further key feature of the ICAP is that the treating therapists (4 Speech and Language Therapists and one Clinical Psychologist) work as a team, meaning all of them will work with each PWA over the 4-week ICAP.

PWA will be grouped into roughly-matched cohorts of 4 (based on aphasia severity). As 'day attenders' they will participate 09:00-17:00 for 4 days a week for 4 weeks, engaging for up to 6 hours a day. Some PWA will travel from home each day. Those who cannot manage this will stay 3 nights a week in a local hotel offering accessible rooms.

The aim is to provide ~100 hours of therapy. The content will involve patient and family education, individual goal-setting, impairment and activity-based therapy (language and communication), conversation-partner training, and facilitative strategies for communication. The interventions will be delivered using a variety of approaches, including individual and paired sessions, group sessions, independent practice (including therapy apps), and sessions with PWA and their family members.

The ICAP will also include a clinical psychology-led forum called Carers' Café to support nominated carers of PWA in adjusting and adapting to the changes they are experiencing. The group will meet weekly and follow the principles of Acceptance and Commitment Therapy [47]. Themes will include 'letting go of the struggle', 'increasing mental flexibility', 'unhooking from the pain and loss', and acknowledging the strain that sometimes accompanies this role. During the ICAP, weekly 1-hour sessions will be held face-to-face where possible, or hybrid if not. The ICAP is an intensive experience for carers and they will need help in providing continued support for the PWA's recovery trajectory after discharge. Accordingly, 4 more weekly remote sessions of Carers' Café will be held following the ICAP to support ongoing adjustment and to establish a legacy of peer support.

Control (standard care) Although the amount of therapy received by PWA in the community varies, the most in-depth study of this variation across 21 UK-based SLT departments concludes as follows: "Where resources are in short supply, therapists have the difficult ethical decision of providing therapeutic levels of intervention to some patients, or providing sub therapeutic levels to all. Currently, it looks as if the latter is most common in practice."[48] This study found the majority of PWA over a year post-stroke were not receiving any therapy, while a minority were receiving ~6.3 hours, ranging widely from 0.5-41.5 hours. To capture the quantity and quality of the therapy received by PWA in this arm (and the ICAP group once they complete the ICAP) we will ensure the research team complete the relevant sections of the Client Service Receipt Inventory at each time point.

DATA MANAGEMENT Confidentiality The study will be managed in compliance with the requirements of the UK General Data Protection Regulation (2021), the UK Data Protection Act (2018), Good Clinical Practice and relevant UCL and NWORTH Standard Operating Procedures. All Investigators and study site staff will comply with the requirements of the UK General Data Protection Regulation (2021) with regards to the collection, storage, processing and disclosure of personal information, and will uphold the Act's core principles. UCL is the data controller; the UCL Data Protection Officer is Spenser Crouch: s.crouch@ucl.ac.uk. The data processors are UCL and NWORTH CTU (Bangor). NWORTH CTU will be holding pseudonymised data and the additional information to identify the pseudonymised data will be held by UCL. The study will be collecting the following personal data: (see data protection registration form)

Data management will be handled by the North Wales Organisation for Randomised Trials in Health CTU with Dr. Zoë Hoare, Principal Statistician and CTU Director, as lead. A study-specific Data Management Plan will be written.

There will be two databases:

1. The participant database held at UCL which will include personalised data, mostly demographics, and clinical data (e.g. name, DoB, region, ethnicity, gender, date of stroke, type of stroke and some behavioural measures)
2. The pseudonymised database held at NWORTH (REDCap) which will contain all the trial data (the baseline and outcome measures which are all behavioural scores). NWORTH will not have access to the identifying information. This will be held at UCL.

ASSESSMENT AND MANAGEMENT OF RISK

Clinical risks (and contingencies):

* Low levels of PWA recruitment. This is unlikely given our previous ICAP was massively oversubscribed despite not advertising the service as we plan to do in this programme. Prof Crinion's aphasia clinic has a backlog of over 100 PWA formally waiting to be assessed for ICAP suitability, with 10 new enquiries per month from clinicians throughout the UK about referrals into the service. With an additional site at St George's and with support from the LCRNs and our charity partners, we are confident we will meet our targets.
* Not collecting data of sufficient quality and quantity to assess current therapy provision in the community for PWA. Our team includes experts who have captured such data previously and we have increased the resources required to collect such data.
* Insufficient variability in terms of time-since-stroke across the study groups. This is unlikely given our previous experience in aphasia assessment clinics at both sites. A discussion of additional risks posed by the intervention and all tests above standard care must be included, and the mitigations of these risks should be detailed in this section. A risk/benefit analysis plus risk management of all interventions involved in the trial should be included.

OVERSIGHT COMMITTEES

Data Monitoring Committee (DMC):

Dr Lotte Meteyard Chair Prof David Howard Member Prof Aidan O'Keeffe Member (external statistician)

Trial Steering Committee (TSC):

Prof Argye Hillis Chair Prof Adam Wagner Member (external statisti1. OVERSIGHT COMMITTEES

Data Monitoring Committee (DMC):

Dr Lotte Meteyard Chair Prof David Howard Member Prof Aidan O'Keeffe Member (external statistican)

Trial Steering Committee (TSC):

Prof Argye Hillis Chair Prof Adam Wagner Member (external statistican) Prof Dorothee Saur Member Ms Becci Haywood Public Member Prof Alex Leff Member

Trial Management Group (TMG) The TMG will include the Chief Investigator and trial staff. The TMG will be responsible for overseeing the trial. The group currently meets monthly.

The TMG will review recruitment figures, SAEs and substantial amendments to the protocol prior to submission to the REC. All PIs will be kept informed of substantial amendments through their nominated responsible individuals.

Other committees The role of the DMC is to provide advice on data and safety aspects of the trial but where not all members are independent. Meetings of the Committee will be held 6 monthly to review interim analyses, or as necessary to address any issues.

can).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years old) PWA caused by stroke
2. More than 3 months post-stroke
3. Can use English to communicate (even if not as their first language)
4. Carers will be nominated (if available) by individual PWA

Exclusion Criteria:

1. Severe speech apraxia (no meaningful spoken word output)
2. Severe fatigue or other reasons they cannot commit to the timing and duration of the ICAP
3. Ongoing debilitating psychiatric disorders (e.g. psychosis, but not low mood)
4. Co-existing neurological disorders affecting engagement (e.g. dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Stroke and Aphasia Quality of Life Scale-39 | Four months post allocation to interventio or control arm.
  The primary outcome measure will be a standardized scale for measuring quality of life for PWA (SAQOL-39g) (44). The primary endpoint is at 4 months, i.e. 3 months post-ICAP. We have a host of secondary measures covering all aspects of WHO ICF (see Flow Diagram). Research assistants blinded to group allocation will collect the outcomes at 4 time points: Baseline, 1-, 4- and 9- months post allocation.
Structural MRI brain scan | Four months post treatment-allocation
  By using a high-resolution MRI brain scan prior to therapy, we will provide a mechanistic account of the effects of the ICAP on PWA's speech production and speech comprehension gains.

SECONDARY OUTCOMES:
Comprehensive Aphasia Test | Baseline, 1-month, 4-month and 9-month post treatment-allocation
  Language impairment
Communicative Effectiveness Index | Baseline, 4-month and 9-month post treatment-allocation
  Functional Communication
Communicative Participation Item Bank | Baseline, 1-month, 4-month and 9-month post treatment-allocation
  Confidence measure
Stroke Aphasic Depression Questionnaire | Baseline, 4-month and 9-month post treatment-allocation
  Measure of mood
General Health Questionnaire-12 | Baseline, 4-month and 9-month post treatment-allocation
  psychological well-being (PWA)
Goal Assessment Scale | Baseline, 1-month, 4-month and 9-month post treatment-allocation
  Short, medium, long-term and economic goals
Client Service Receipt Inventory | Baseline, 1-month, 4-month and 9-month post treatment-allocation
  Utilization of health, social, and community services
Adult Carers Quality Of Life Questionnaire | Baseline, 4-month and 9-month post treatment-allocation
  Carer quality of life
Zarit Burden Interview | Baseline, 4-month and 9-month post treatment-allocation
  Carer burden
Patient Health Questionnaire-9 | Baseline, 4-month and 9-month post treatment-allocation
  Psychological well-being

OTHER OUTCOMES:
Qualitative interviews | 9-months
  With both PWA and carers

CONTACTS AND LOCATIONS:
Locations (1):
- UCL Queen Square Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised data set will be made available for other researchers to request access to for perpetuity.